CLINICAL TRIAL: NCT05582668
Title: Sarcopenia After Bariatric Surgery in Older Patients: a Cohort Study
Acronym: SABO
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S66815
Record Dates: First submitted 2022-10-12; First posted 2022-10-17 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2024-10

CONDITIONS: Overweight and Obesity; Bariatric Surgery; Aging; Sarcopenic Obesity
MeSH Terms: conditions — Overweight; Obesity | interventions — Bariatric Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Cohort 1: Cohort 1: Older patients with overweight, obesity after bariatric surgery
  Interventions: Procedure: Bariatric surgery
- Cohort 2: Cohort 2: Older patients with overweight, obesity without bariatric surgery

INTERVENTIONS:
Procedure: Bariatric surgery — Bariatric surgery
  Groups: Cohort 1

SUMMARY:
The retrospective cohort study will compare the prevalence of sarcopenia and associated factors between older patients who have undergone bariatric surgery and older patients with obesity without previous bariatric surgery.

DETAILED DESCRIPTION:
The aim of the study is to compare the prevalence of sarcopenia and nutritional status between adults older than 65 years who have previously undergone bariatric surgery and patients with obesity but without previous bariatric surgery. Current sarcopenia will be assessed during a cross-sectional assessment after surgery using the criteria from the European Working Group on Sarcopenia in Older People (EWGSOP).

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Age 65 years or older
* Cohort 1 (exposed): Previous bariatric surgery for obesity at least 1 one year ago
* Cohort 2 (unexposed): No previous weight loss surgery

Exclusion Criteria:

* Current diagnosis of cancer
* Advanced organ failure, including chronic kidney disease Stage 5, liver cirrhosis Stage 3, intestinal failure, heart failure stage D, or chronic obstructive pulmonary disease stage 4.
* Immobility
* Neuromuscular degenerative conditions

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Subjects with overweight, obesity or after bariatric surgery
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2022-10-03 (Actual); Primary Completion 2024-07-14 (Actual); Study Completion 2024-07-14 (Actual)

PRIMARY OUTCOMES:
The number of older patients with sarcopenia after bariatric surgery compared to non-surgical control patients. | At least one year post surgery
  a) Sarcopenia will be classified according to the criteria form the European Working Group on Sarcopenia in Older People revised guidelines (EWGSOP2) based on skeletal muscle mass, muscle strength and physical performance criteria.

SECONDARY OUTCOMES:
1. Appendicular skeletal muscle mass older of patients after bariatric surgery compared to non-surgical control patients | At least one year post surgery
  1. Appendicular skeletal muscle mass older of patients after bariatric surgery compared to non-surgical control patients
2. The prevalence of nutrient deficiencies in older patients after bariatric surgery compared to non-surgical control patients. | At least one year post surgery
  a. Indices of nutrient deficiencies will include reported dietary intake of protein, zinc, selenium, and blood levels of Vitamin D, zinc, and selenium.
3. Markers of chronic systemic inflammation in older patients after bariatric surgery compared to non-surgical control patients | At least one year post surgery
  Inflammatory markers will include CRP, IL-1β, IL-6, IL-8, TNF-α

CONTACTS AND LOCATIONS:
Locations (1):
- Obesity Clinic University Hospitals Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Eksteen G, Vanuytsel T, Vangoitsenhoven R, Mertens A, Lannoo M, De Leus E, Van der Schueren B, Matthys C. Sarcopenia, Muscle Mass and Protein Intake in Adults Older Than 65 Years After Earlier Bariatric Surgery. J Cachexia Sarcopenia Muscle. 2025 Jun;16(3):e13839. doi: 10.1002/jcsm.13839. PMID 40468919